CLINICAL TRIAL: NCT05762133
Title: African-American Social Support Effectiveness Treatment-Partners Alleviating Perinatal Depression
Brief Title: African-American Social Support Effectiveness Treatment
Acronym: ASSET-PPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Sheehan David Fisher, Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1R21MD014798-01A1 (NIH)
Record Dates: First submitted 2023-02-27; First posted 2023-03-09 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Maternal Perinatal Depression
Keywords: perinatal depression; postpartum depression; anxiety; fathers; partners; parents; African American; social support
MeSH Terms: conditions — Depression, Postpartum; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: We plan to enroll 50 parent dyads (100 individuals total, 25 romantic or non-romantic partners per arm). If we assume 5% attrition at each phase, we anticipate analyzable data for between 20-25 parent duos per arm.
Who Masked: Outcomes Assessor
Masking Description: At 3- and 6-months postpartum, mothers and fathers will attend an observation that includes a 5-minute free play with their infant separately and a 5-minute free play together as co-parents. Parent-infant interactions will be videotaped and interaction quality will be coded by a blind evaluator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ASSET-PPD intervention group (Experimental): 25 parent dyads with a mother who is receiving individual treatment outside of the study and the father is receiving the ASSET-PPD training
  Interventions: Behavioral: African-American Social Support Effectiveness Treatment-Partners alleviating Perinatal Depression (ASSET-PPD)
- No additional treatment group (No Intervention): 25 parent dyads with a mother who is receiving individual treatment outside of the study and the father is not receiving the ASSET-PPD training

INTERVENTIONS:
Behavioral: African-American Social Support Effectiveness Treatment-Partners alleviating Perinatal Depression (ASSET-PPD) — This proposed novel intervention has four prenatal modules and two postpartum review sessions addressing key correlates of Perinatal Depression (PND) with the largest effect sizes by targeting fathers': 1) prenatal and postpartum family involvement; 2) mental health psychoeducation; 3) interparental communication and relationship skills; and 4) balanced division of family tasks. The intervention is based on the stress-generation and cognitive-behavior theories to frame skill-based individual sessions of didactics, interactive training, and trackable objectives.
  Arms: ASSET-PPD intervention group

SUMMARY:
The objective of this treatment study is to develop and test an augmentation therapy in conjunction with maternal psychiatric treatment that targets the fathers' support of the mothers' mental health and contributions to the family environment to reduce maternal stress. The African-American Social Support Effectiveness Treatment-Partners alleviating Perinatal Depression (ASSET-PPD) intervention will be delivered to fathers in an individual setting to target the context in which a mother lives to expand her support beyond the direct reach of her treatment professional. This study provides skills and training to fathers who have a partner with prenatal depression. The aim is to reduce maternal depression during the perinatal period and improve the family environment for the infant.

DETAILED DESCRIPTION:
African-American (AA) mothers have a higher risk for perinatal depression than Caucasian women that is attributable to increased socio-environmental stressors. In addition, AA women have poor healthcare utilization and compliance with psychiatric treatment compared to Caucasian women. An intervention is required to supplement and support the clinical objectives of the mother's depression care without requiring the mother's direct involvement. Fathers are an underutilized resource to reduce the mother's environmental stress and encourage healthy maternal behaviors. The African-American Social Support Effectiveness Treatment- Partners alleviating Perinatal Depression (ASSET-PPD) protocol will target the fathers' support of the mothers' mental health treatment and their active engagement in the family to reduce maternal stress. The ASSET-PPD intervention will be designed to have 4 active modules that address key factors to reduce maternal stress during the prenatal period and 2 postpartum review sessions. The modules will be individual sessions constructed to provide training, information, and behavioral assignments to increase fathers': 1) prenatal and postpartum family involvement; 2) mental health psychoeducation; 3) interparental communication and relationship skills; and 4) balanced division of family tasks. ASSET-PPD will be evaluated in a pilot Randomized Clinical Trial (RCT) with 50 cohabitating or non-cohabitating fathers and AA mothers who will be randomized into the ASSET-PPD intervention or the comparator group. Fathers only will participate in the intervention, and mothers and fathers will complete measures of mental health and parental experiences. Maternal depressive symptoms will be assessed as a primary outcome, and breastfeeding and parent-infant interactions will be assessed as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Parents will be 18 years of age or older.
* Parents are eligible for the study if the woman is in the 2nd trimester, she is receiving psychiatric treatment for depression with a score of 11 or greater on the Inventory of Depressive Symptoms-Self-Rated (IDS-SR16), which indicates clinically significant symptoms, and the mother is African-American
* Parents do not need to be romantic partners to be eligible. Infants (0-6 months) are included in the study to examine the parent-infant interactions

Exclusion Criteria:

The parents will be excluded if:

* There is report of ongoing physical or sexual abuse
* They have plans to terminate the pregnancy
* The woman is showing symptoms of hypomania/mania, psychosis, or substance use in the past 12 months

Father will be excluded if he:

* Has symptoms of psychosis in the past 12 months
* Has below 6th grade education
* Has difficulty focusing on 1 hour of instruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligibility for this study includes parent dyads of female-male co-parents.
Enrollment: 100 (Actual)
Dates: Start 2020-08-27 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Maternal depression | Second trimester through six month postpartum
  The Inventory of Depressive Symptoms-Self-Rated (IDS-SR16) is a 16-item self-report measure of depressive symptoms. Minimum value: 0, Maximum value: 3, Higher scores indicate worse outcome
Maternal anxiety | Second trimester through six month postpartum
  The Generalized Anxiety Disorder-7-item (GAD-7) is a 7-item, self-report measure assesses the dimension of generalized anxiety. Minimum value: 0, Maximum value: 3, Higher scores indicate worse outcome

SECONDARY OUTCOMES:
Breastfeeding | Administered at 1-, 3-, and 6-months
  The FeedCat Tool (FT) is a 9-item self-report breastfeeding assessment that measures the type, amount, and mode of feeding. FT complies with the World Health Organization (WHO) and Centers for Disease Control (CDC) recommendations
Infant affect and mood regulation | Administered at 1-, 3-, and 6-months
  The Infant Behavior Questionnaire- Revised (IBQ-R) is a 36-item parent-report measure of infant behaviors (positive/negative affect, regulation), Minimum value: 0, Maximum value: 7, Higher scores indicate greater level of temperament dimension of the 14 scales
Parent-infant interaction quality | At 3- and 6-months
  Mothers and fathers will attend an onsite observation that includes a 5-minute free play with their infant separately and a 5-minute free play together as co-parents. Parent-infant interactions will be videotaped by a split-screen Noldus Media Recorder. Interaction quality will be coded on the Parent-Child Early Relational Assessment (PCERA). PCERA is a valid, reliable measure of the quality of affect and behavior in parent-child interactions and has been used in psychiatric studies and triadic interactions. Minimum value: 1, Maximum value: 5, Higher scores indicate better outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No